CLINICAL TRIAL: NCT06790043
Title: Randomized Control Trial: Impact of Patient Selected Visual Art in the Hospital Room During Antepartum Admission on Hospital Satisfaction Scores and Patient Experience.
Brief Title: Impact of Patient Selected Visual Art in the Hospital Room During Antepartum Admission on Hospital Satisfaction Scores and Patient Experience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6960
Record Dates: First submitted 2024-12-11; First posted 2025-01-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Pregnancy Complications; Hospital Environment; Hospitalization; Satisfaction, Patient
Keywords: Visual Art; Antepartum Hospitalization
MeSH Terms: conditions — Pregnancy Complications; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual art Intervention (Experimental): Patient-selected visual art Routine care
  Interventions: Other: Patient-selected visual art in hospital room
- Control (Active Comparator): Routine care
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Patient-selected visual art in hospital room — Patient-selected visual art placed in patient's antepartum hospital room
  Other Names: Patient-selected visual art; Visual art
  Arms: Visual art Intervention
Other: Routine care — Patient will receive routine care, and will not select, nor have, visual art in their antepartum hospital room.
  Other Names: Control; No visual art
  Arms: Control

SUMMARY:
The purpose of this study is to assess whether patient-selected visual art for patients admitted to the antepartum unit will increase hospital satisfaction compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* patients who are greater than or equal to 18 years of age
* patients admitted to the study hospital's antepartum unit for care
* currently pregnant
* willing and able to provide informed consent and complete the provided questionnaire

Exclusion Criteria:

* patients less than 18 years of age
* patients who are not pregnant
* patients who are not admitted to study hospital's antepartum unit
* patients who cannot provide informed consent in English
* patients who have participated in this study during a previous admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HCAHPS Survey Overall Hospital Rating | through study completion, an average of 2 years
  Overall hospital rating question #18 from HCAPHS Survey

SECONDARY OUTCOMES:
Qualitative Experience | through study completion, an average of 2 years
  Likert Scale Questions and Open-ended Questions regarding patient's experience with visual art and hospital stay
Portion of HCAHPS Survey regarding Patient Experience | through study completion, an average of 2 years
  Likert and Rating of patient's experience of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dexter, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lankston L, Cusack P, Fremantle C, Isles C. Visual art in hospitals: case studies and review of the evidence. J R Soc Med. 2010 Dec;103(12):490-9. doi: 10.1258/jrsm.2010.100256. PMID 21127332
- [Background] George DR, Boer C, Hammer J, Hopkins M, King T, Green MJ. Evaluating the Benefits of Hospital Room Artwork for Patients Receiving Cancer Treatment: A Randomized Controlled Trial. J Hosp Med. 2018 Aug 1;13(8):558-561. doi: 10.12788/jhm.2915. Epub 2018 Feb 5. PMID 29401210
- [Background] Monsuez JJ, Francois V, Ratiney R, Trinchet I, Polomeni P, Sebbane G, Muller S, Litout M, Castagno C, Frandji D. Museum Moving to Inpatients: Le Louvre a l'Hopital. Int J Environ Res Public Health. 2019 Jan 13;16(2):206. doi: 10.3390/ijerph16020206. PMID 30642107
- [Background] Karnik M, Printz B, Finkel J. A Hospital's Contemporary Art Collection: Effects on Patient Mood, Stress, Comfort, and Expectations. HERD. 2014 Spring;7(3):60-77. doi: 10.1177/193758671400700305. PMID 24782236
- [Background] Crane T, Buultjens M, Fenner P. Art-based interventions during pregnancy to support women's wellbeing: An integrative review. Women Birth. 2021 Jul;34(4):325-334. doi: 10.1016/j.wombi.2020.08.009. Epub 2020 Sep 8. PMID 32912739
- [Background] Eminovic S, Vincze G, Fink A, Fischerauer SF, Sadoghi P, Leithner A, Kamolz LP, Tscheliessnigg K, Bernhardt GA. Positive effect of colors and art in patient rooms on patient recovery after total hip or knee arthroplasty : A randomized controlled trial. Wien Klin Wochenschr. 2022 Mar;134(5-6):221-226. doi: 10.1007/s00508-021-01936-6. Epub 2021 Sep 7. PMID 34491443
- [Background] Iyendo TO, Uwajeh PC, Ikenna ES. The therapeutic impacts of environmental design interventions on wellness in clinical settings: A narrative review. Complement Ther Clin Pract. 2016 Aug;24:174-88. doi: 10.1016/j.ctcp.2016.06.008. Epub 2016 Jul 1. PMID 27502819